CLINICAL TRIAL: NCT04143360
Title: Improvement and Clinical Application of a New Minimally Invasive Closed Thoracic Drainage System
Brief Title: Improvement and Application of New Closed Drainage Device
Acronym: IAAONCDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yongxin Zhou (Other)
Responsible Party: Sponsor-Investigator, Yongxin Zhou, Director, Shanghai Tongji Hospital, Tongji University School of Medicine
Organization: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-LCYJ-012
Record Dates: First submitted 2019-09-29; First posted 2019-10-29 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Hydrothorax; Pneumothorax
MeSH Terms: conditions — Hydrothorax; Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Closed Drainage Device (Experimental): We further improve the new closed thoracic drainage system by changing the material of drainage tube, adding external fixator control valve and increasing the gas flow monitoring kit for special patients, and apply it in clinical practice.
  Interventions: Device: New Closed Drainage Device
- Traditional Closed Drainage Device (Experimental): We use traditional closed drainage devices for patients with hemothorax and pneumothorax.
  Interventions: Device: Traditional closed drainage device

INTERVENTIONS:
Device: New Closed Drainage Device — For the first group, a new closed drainage device was adopted.
  Arms: New Closed Drainage Device
Device: Traditional closed drainage device — For group 2, conventional closed drainage device was used.
  Arms: Traditional Closed Drainage Device

SUMMARY:
According to the problems of traditional closed thoracic drainage in clinical work, this study aims to further improve and improve the new closed thoracic drainage system by changing the material of drainage tube, increasing the regulating valve of external fixator and increasing the gas flow monitoring kit for special patients, so as to expand its clinical application scope and formulate its operation. Standardize. At the same time, through a randomized controlled study, the simplicity, effectiveness and safety of the new minimally invasive thoracic closed drainage system developed by the research group were deeply studied.

DETAILED DESCRIPTION:
The traditional closed thoracic drainage method has complex operation and high technical requirements. It has obvious pain during and after operation. Operational complications such as tissue organs, intercostal vessels and nerve injury may occur during the operation. Accidents may also occur after catheterization, including leakage around thoracic drainage tube, thoracic drainage tube prolapse, subcutaneous emphysema and accumulation. Liquid; To solve these problems, we have invented "minimally invasive thoracic closed drainage system" through a number of patent designs, including: thoracic closed drainage tube implantation expansion forceps, double-chamber thoracic drainage device with side balloon, guide wire, puncture needle, various types of dilators, chest tube fixation devices, etc. The system has the characteristics of minimally invasive puncture and implantation of drainage tube, safe, fast operation, no need of suture and fixation, good position of drainage tube after implantation, less pain for patients, and closing incision in the medial part of patients, avoiding leakage and subcutaneous emphysema and hydrops.

ELIGIBILITY:
The selection criteria were as follows:

* age 18-70 years, gender is not limited;
* subjects clearly understand the purpose of the study, are willing and able to comply with the requirements to complete the study and sign the informed consent;
* 18 Kg/m2 < BMI < 25 Kg/m2;
* patients who need thoracic closed drainage for exhaust and drainage because of pneumothorax volume > 30%;
* subjects did not have serious chest wall deformities.

Exclusion criteria:

* Patients at high risk of bleeding, including patients with congenital hemophilia, thrombocytopenia (PLT < 50 *109/L), platelet dysfunction (such as idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, congenital platelet dysfunction);
* Cardiopulmonary function is poor, which is not suitable for the participants.
* Patients with other infectious diseases (inflammation, tuberculosis) or empyema in the thoracic cavity;
* Infection of skin around puncture and drainage;
* Participated in other clinical trials within 30 days;
* Other reasons why the researchers think it is inappropriate to participate in the experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Total drainage time | up to 24 weeks
  Efficiency of treatment
Pulmonary reexpansion ratio | up to 24 weeks
  Pulmonary reexpansion ratio

SECONDARY OUTCOMES:
VAS pain score during and after operation | up to 24 weeks
  0 points means no pain; 1 points - 3 points means mild pain that patients can tolerate; 4 points - 6 points means pain affect sleep, but patients can tolerate;7 points - 10 points: means patients have gradually strong pain, which have affected appetite and sleep.

OTHER OUTCOMES:
Operation time of thoracentesis | up to 24 hours
  Operation time of thoracentesis
Percentage of lung recruitment on day 1 and 3 | up to 24 weeks
  Percentage of lung recruitment
Operational-related complications | up to 24 weeks
  Incidence of loss of thoracic wall nerves, intercostal vessels and thoracic and abdominal organs
Incidence of related accidents after catheterization | up to 24 weeks
  Incidence rate of peri-drainage tube exudation, drainage tube falling off, drainage tube obstruction and subcutaneous emphysema
The size of the wound | up to 24 weeks
  The size of the wound
infection of the wound | up to 24 weeks
  infection of the wound

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang WP, Ni YF, Wei YN, Li XF, Cheng QS, Lu Q. Bronchiolitis obliterans complicating a pneumothorax after Stevens-Johnson syndrome induced by lamotrigine. J Formos Med Assoc. 2015 Mar;114(3):285-9. doi: 10.1016/j.jfma.2012.02.026. Epub 2012 Jun 6. PMID 25777978
- [Result] Khan BA, Reddy PM, Khan AM. Spontaneous pneumothorax in the immediate post-operative hour in a primigravida following emergency caesarean section under spinal anaesthesia. Indian J Anaesth. 2015 Feb;59(2):126-9. doi: 10.4103/0019-5049.151380. No abstract available. PMID 25788749
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=Bronchiolitis+obliterans+complicating+a+poeumothorax+after+Stevens-+Johson+syndrome+induced+by+lamotrigine.
- See also: pubmed — http://www.ncbi.nlm.nih.gov/pubmed/?term=Spontaneous+pneumothorax+in+the+immediate+post-operative+hour+in+a+primigravida+following+emergency+caesarean+section+under+spinal+anaesthesia.